CLINICAL TRIAL: NCT00611247
Title: Phase II Study of Two Distinct Tailored Temozolomide Regimens for Patients With Acute Myeloid Leukemia Age > 60 Years and Poor Risk/Refractory Disease
Brief Title: Phase 2 Study of Temozolomide to Treat Poor Risk / Refractory Acute Myeloid Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bruno C. Medeiros (Other)
Collaborators: Schering-Plough (Industry)
Responsible Party: Sponsor-Investigator, Bruno C. Medeiros, PI, Stanford University
Organization: Stanford University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-07815; 97611 (Other: Stanford University Alternate IRB Approval Number); SU-12142007-936 (Other: Stanford University); HEMAML0004 (Other: OnCore); NCT00426309 (obsolete NCT alias)
Record Dates: First submitted 2008-01-25; First posted 2008-02-08 (Estimated); Results first posted 2014-07-09 (Estimated); Last update posted 2018-06-15 (Actual); Status verified 2018-05

CONDITIONS: Leukemia, Myeloid
MeSH Terms: conditions — Leukemia, Myeloid | interventions — Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Methylated AGAT Promoter (Group 1) (Experimental): Induction: 200 mg/m2/day oral Temozolomide x 7 days
  Interventions: Drug: Temozolomide
- Un-Methylated AGAT Promoter (Group 2) (Experimental): Priming: 100 mg/m2/day oral Temozolomide x 14 days, followed by Induction: 200 mg/m2/day oral Temozolomide x 7 days
  Interventions: Drug: Temozolomide

INTERVENTIONS:
Drug: Temozolomide — Priming, Group 2 only, 100 mg/m2/day temozolomide.
  Induction (both arms) 200 mg/m2/day temozolomide
  Other Names: Temodar, Temodal

SUMMARY:
Open-label, non-randomized, parallel assignment, phase 2 trial assessing the safety and efficacy of distinct temozolomide treatment regimens for patients with AML and poor prognosis

DETAILED DESCRIPTION:
This is a single institution phase 2 clinical trial evaluating the efficacy, safety, and tolerability of tailored temozolomide therapy for patients with acute myeloid leukemia (AML) and poor risk features.

Patients will be assigned to 1 of 2 parallel treatment groups based on their AGAT promoter region methylation status, as determined by PCR.

Patients achieving a complete remission after 1 to 2 cycles of chemotherapy will be eligible to receive up to an additional 5 cycles of temozolomide of 5 or 19 days, depending on the methylation status of the AGAT promoter (consolidation phase).

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically or cytologically confirmed Acute Myeloid Leukemia, as defined by the WHO classification.
2. Patients must be considered unfit for conventional induction chemotherapy, unwilling to receive such treatment or have evidence of disease relapse or refractory disease.
3. For patients who have received no prior conventional chemotherapy, one of the following must be present:

   * Poor risk cytogenetics (complex abnormalities, deletions of chromosome 7 or 5, 11q23 abnormalities, inv[3])
   * Secondary leukemia (prior hematologic disorder or therapy-related leukemia).
4. Age > 60 years of age.
5. Life expectancy of greater than 3 months.
6. ECOG performance status greater than 2.
7. Patients must have normal organ and marrow function as defined below:
8. Adequate hepatic function: Total bilirubin 1.5mg/dL, AST(SGOT)/ALT(SGPT) 2.5 X institutional upper limit of normal.
9. Adequate renal function: serum creatinine within normal institutional limits or Calculated creatinine clearance > 60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal.
10. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier.
2. Patients may not be receiving any other investigational agents.
3. History of allergic reactions attributed to compounds of similar chemical or biologic composition to temozolomide or DTIC
4. History of gastrointestinal disease or significant bowel resection that could interfere with drug absorption.
5. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
6. Prior allogeneic stem cell transplantation.
7. Inability to swallow tablets
8. Prior radiation up to more than 25% of bone marrow.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2007-12; Primary Completion 2009-12 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Carneiro de Medeiros, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

REFERENCES:
- [Result] Medeiros BC, Kohrt HE, Gotlib J, Coutre SE, Zhang B, Arber DA, Zehnder JL. Tailored temozolomide therapy according to MGMT methylation status for elderly patients with acute myeloid leukemia. Am J Hematol. 2012 Jan;87(1):45-50. doi: 10.1002/ajh.22191. Epub 2011 Nov 4. PMID 22052619
- [Result] Bruno C Medeiros, Holbrook E Kohrt, Richa Rajwanshi, Jason Gotlib, Steven E Coutre, Michaela Liedtke, Caroline Berube, Melody Zhang, Daniel A Arber, James L Zehnder. "Temozolomide In Acute Myeloid Leukemia: A MGMT Promoter Methylation Status-Based Treatment Stratification." Blood. 2010;116(21) (abs 3313).

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 42 subjects consented to screening for this study.
Pre-assignment Details: 6 of 42 subjects did not meet eligibility criteria and did not receive induction therapy. Of these, 1 subject had no evidence of AML; 1 had acute lymphoblastic leukemia, and 4 had disease progression and death before induction. None of the 6 were stratified to a treatment group, and were not treated on study.
Period: Overall Study
Arm/Group | Methylated AGAT Promoter (Group 1) | Un-Methylated AGAT Promoter (Group 2)
Started | 5 | 31
Completed | 3 | 10
Not Completed | 2 | 21
Not completed — Death | 1 | 5
Not completed — Lack of Efficacy | 1 | 16

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Methylated AGAT Promoter (Group 1) | Un-Methylated AGAT Promoter (Group 2) | Total
Number analyzed (Participants) | 5 | 31 | 36
Age, Continuous [Median (Full Range); unit: years] | 77 [66 to 83] | 75 [64 to 87] | 75 [64 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 11 | 13
  Male | 3 | 20 | 23

OUTCOME MEASURES:

1. Primary Outcome: Response Rate (CR + CRi + LFS)
Description: Response determined per European LeukemiaNet response criteria:
  CR = bone marrow blasts <5%; absence of blasts with Auer rods; absence of extramedullary disease; absolute neutrophil count > 1.0 x 10e9/L; platelet count > 100 x 10e9/L; and independence of red cell transfusions.
  CRi = all CR criteria except for residual neutropenia (< 1.0 x 10e9/L) or thrombocytopenia (< 100 x 10e9/L)].
  Morphologic leukemia-free state (LFS) = bone marrow blasts <5%; absence of blasts with Auer rods; absence of extramedullary disease; with no hematologic recovery required.
  Relapse = bone marrow blasts >5%; reappearance of blasts in the blood; or development of extramedullary disease.
Time Frame: up to 2 months
Measure: Number; unit: participants
Arm/Group | Methylated AGAT Promoter (Group 1) | Un-Methylated AGAT Promoter (Group 2)
Number analyzed (Participants) | 5 | 31
participants | 3 | 10

2. Secondary Outcome: Toxicity Profile: Total Number of Drug-related Serious Adverse Events
Time Frame: 12 months
Measure: Number; unit: events
Groups:
- Un-Methylated AGAT Promoter (Group 2): Priming: 100 mg/m2/day oral Temozolomide x 14 days, then followed by Induction: 200 mg/m2/day oral Temozolomide x 7 days
Arm/Group | Methylated AGAT Promoter (Group 1) | Un-Methylated AGAT Promoter (Group 2)
Number analyzed (Participants) | 5 | 31
events | 4 | 27

3. Secondary Outcome: Toxicity Profile: Individual Subjects With Drug-related SAEs
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | Methylated AGAT Promoter (Group 1) | Un-Methylated AGAT Promoter (Group 2)
Number analyzed (Participants) | 5 | 31
participants | 4 | 13

ADVERSE EVENTS:
Arm/Group | Methylated AGAT Promoter (Group 1) | Un-Methylated AGAT Promoter (Group 2)
Serious Adverse Events (participants affected / at risk) | 4/5 | 28/31
Other Adverse Events (participants affected / at risk) | 3/5 | 23/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Methylated AGAT Promoter (Group 1) (N=5) | Un-Methylated AGAT Promoter (Group 2) (N=31)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 4 (5) | 13 (21)
Blood and lymphatic system disorders - Other, Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Arthralgia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Multi-organ failure (General disorders) | 0 (0) | 1 (1)
Sudden death NOS (General disorders) | 0 (0) | 2 (2)
Death NOS (General disorders) | 1 (1) | 3 (3)
Mucosa infection (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Creatinine increased (Investigations) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 1 (2) | 10 (14)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Urinary tract infection (Renal and urinary disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, fever/pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, Multilobar pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Hypoalbuminemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Oral Pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (3) | 12 (17)
White blood cell decreased (Investigations) | 1 (3) | 6 (6)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Methylated AGAT Promoter (Group 1) (N=5) | Un-Methylated AGAT Promoter (Group 2) (N=31)
Anemia (Blood and lymphatic system disorders) | 2 (5) | 19 (36)
Blood and lymphatic system disorders - Not otherwise specified (Blood and lymphatic system disorders) | 1 (1) | 1 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 3 (3)
Lymph node pain (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hemolysis (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 2 (2)
Cardiac disorders - Not otherwise specified (Cardiac disorders) | 1 (1) | 1 (1)
Eye disorders - Not otherwise specified (Eye disorders) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 3 (4)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 5 (8)
Constipation (Gastrointestinal disorders) | 0 (0) | 8 (11)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 6 (7)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 3 (3)
Nausea (Gastrointestinal disorders) | 0 (0) | 10 (13)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2)
Rectal Pain (Gastrointestinal disorders) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 5 (7)
Edema limbs (General disorders) | 0 (0) | 6 (11)
Fatigue (General disorders) | 3 (7) | 19 (24)
Fever (General disorders) | 1 (3) | 2 (2)
Localized edema (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 3 (4)
Lip infection (Infections and infestations) | 1 (1) | 0 (0)
Infections and infestations - Not otherwise specified (Infections and infestations) | 0 (0) | 4 (5)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Activated partial thromboplastin time prolonged (Investigations) | 1 (2) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 4 (7)
Alkaline phosphatase increased (Investigations) | 1 (2) | 4 (4)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0)
Creatinine increased (Investigations) | 2 (4) | 8 (11)
Neutrophil count decreased (Investigations) | 1 (1) | 3 (7)
Platelet count decreased (Investigations) | 1 (2) | 13 (19)
Weight loss (Investigations) | 1 (1) | 4 (4)
White blood cell decreased (Investigations) | 1 (2) | 9 (19)
Anorexia (Metabolism and nutrition disorders) | 1 (2) | 8 (9)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (5) | 13 (18)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (4) | 10 (17)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (2) | 5 (5)
Hypokalemia (Metabolism and nutrition disorders) | 1 (4) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 1 (2) | 7 (9)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Dizziness (Nervous system disorders) | 0 (0) | 3 (3)
Memory impairment (Nervous system disorders) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 1 (2) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Confusion (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 3 (3)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (3)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 3 (3)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 2 (2)
Vaginal hemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 6 (6)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 3 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (3)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (5)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 5 (5)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Hypertension (Vascular disorders) | 0 (0) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No